CLINICAL TRIAL: NCT04804852
Title: Assessment of the Prevalence of Sarcopenia by CT Scan in Patients Diagnosed With Head & Neck Carcinoma
Brief Title: Assessment of the Prevalence of Sarcopenia by CT Scan in Patients Diagnosed With Head & Neck Cancer
Acronym: SARVADS 1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Weprom (Other)
Responsible Party: Sponsor
Other Study IDs: WP-2020-04
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-03

CONDITIONS: Sarcopenia; Cancer of Head and Neck; CT Scan
MeSH Terms: conditions — Sarcopenia; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study population: Patient diagnosed with head & neck carcinoma at diagnosis
  Interventions: Other: sarcopenia assessment

INTERVENTIONS:
Other: sarcopenia assessment — evaluation of sarcopenia by CT san at the C3 vertebrae

SUMMARY:
Sarcopenia is defined by the reduction in skeletal muscle mass and physical performance. It results in a decrease in muscle strength, overall physical activity, walking and the development of balance disorders and falls. It is one of the natural consequences of aging and contributes to frailty and the appearance of geriatric syndrome (s) (Chandapasirt et al, 2015; Cruz-Jentoft et al, 2010).

Its prevalence in patients with Head & Neck cancer is 39% (Hua et al, 2020) and is associated with an increase in postoperative complications (Achim et al, 2017; Bril et al, 2019), with greater toxicity of chemotherapy. (Wendrich et al, 2017) and reduced overall survival (Hua et al, 2020).

It is measured by CT scan (assessment of muscle volume with respect to L3 using IMAGE J software) (Teigen et al, 2018) and by clinical tests (performance tests) (Swartz et al, 2016, Cruz-Jentoft et al, 2010).

Several studies have shown a possible assessment of sarcopenia by measuring skeletal muscle mass with regard to C3 (Ufuk et al, 2019; Swartz et al, 2016).

This trial aims to evaluate the prevalence of sarcopenia in head and neck cancer evaluated by CT at C3.

ELIGIBILITY:
Inclusion Criteria:

* patient over 18 years old,
* affiliated to the social security scheme,
* suffering from locally advanced head & neck cancer (stages I to IVB) at diagnosis,
* not operable,
* justifying treatment by radiotherapy, whether or not associated with chemotherapy or targeted therapy (eg: monoclonal antibodies, immunotherapy) whatever the proposed modalities.

Exclusion Criteria:

* patient treated by non-conservative surgery and cervical lymph node dissection making it impossible to assess muscle mass with regard to C3,
* metastatic disease,
* minor patient,
* adult patient under guardianship,
* pregnancy or breastfeeding in progress.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patient diagnosed with head & neck carcinoma non operable and treated by radiotherapy and/or chemotherapy and/or targeted therapy.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of the prevalence of sarcopenia by cervical CT scan (C3) | 6 months
  Number of patients with sarcopenia at diagnosis and during treatments

SECONDARY OUTCOMES:
Assessment of hypoalbuminemia | 6 month
  Number of patients presenting an hypoalbuminemia.
De- and undernutrition | 6 month
  Number of patients with a BMI <18 and with a prescription for nutritional complements.
Compliance to the treatment | 6 months
  Number of patients having the complete planned treatment
complete response rate | 6 months
  Number of patients with a complete response on the end-of-treatment evaluation scanner according to the RECIST or PERCIST criteria in the numerator out of the total number of patients in the denominator
Assessment of hospitalizations treatment-related complications | 6 months
  Number of hospitalizations per patient for treatment-related complications

CONTACTS AND LOCATIONS:
Overall Officials: LE DU Katell, MD, Study Director — Weprom
Locations (1):
- Clinique Victor Hugo / Centre Jean Bernard, Le Mans, France

IPD SHARING:
Plan to Share IPD: No